CLINICAL TRIAL: NCT06252649
Title: Phase 3 Multicenter, Randomized, Open-label, Active-controlled Study of Sotorasib, Panitumumab and FOLFIRI Versus FOLFIRI With or Without Bevacizumab-awwb for Treatment-naïve Subjects With Metastatic Colorectal Cancer With KRAS p.G12C Mutation (CodeBreaK 301)
Brief Title: Study of Sotorasib, Panitumumab and FOLFIRI Versus FOLFIRI With or Without Bevacizumab-awwb in Treatment-naïve Participants With Metastatic Colorectal Cancer With KRAS p.G12C Mutation
Acronym: CodeBreaK 301
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210081
Record Dates: First submitted 2024-01-15; First posted 2024-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Sotorasib; Panitumumab; FOLFIRI; Bevacizumab-awwb; Oncology
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — sotorasib; Panitumumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Sotorasib + Panitumumab + FOLFIRI (Experimental): Sotorasib will be taken daily (QD) as an oral tablet. Panitumumab and FOLFIRI will be received every 2 weeks (Q2W) via intravenous (IV) infusion.
  Interventions: Drug: FOLFIRI Regimen; Drug: Sotorasib; Drug: Panitumumab
- Arm B: FOLFIRI with or Without Bevacizumab-awwb (Active Comparator): Participants will receive FOLFIRI Q2W with or without bevacizumab-awwb.
  Interventions: Drug: FOLFIRI Regimen; Drug: Bevacizumab-awwb

INTERVENTIONS:
Drug: FOLFIRI Regimen — Combination of irinotecan, leucovorin, and 5-fluorouracil given via IV infusion Q2W.
Drug: Sotorasib — Immediate-release solid dosage form administered orally.
  Other Names: AMG 510; Lumakras; Lumykras
  Arms: Arm A: Sotorasib + Panitumumab + FOLFIRI
Drug: Panitumumab — Administered via IV infusion Q2W.
  Other Names: Vectibix
  Arms: Arm A: Sotorasib + Panitumumab + FOLFIRI
Drug: Bevacizumab-awwb — Administered via IV infusion Q2W.
  Other Names: MVASI
  Arms: Arm B: FOLFIRI with or Without Bevacizumab-awwb

SUMMARY:
The aim of this study is to compare progression free survival (PFS) in treatment-naïve participants with KRAS p.G12C mutated metastatic colorectal cancer (mCRC) receiving sotorasib, panitumumab and FOLFIRI vs FOLFIRI with or without bevacizumab-awwb.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented metastatic colorectal adenocarcinoma with KRAS p.G12C mutation by a locally validated assay.
* Central laboratory detection of KRAS p.G12C mutation.
* Measurable metastatic disease per RECIST v1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1.
* Adequate organ function.

Exclusion Criteria:

* Active, untreated brain metastases.
* Leptomeningeal disease
* Previous treatment with a KRAS p.G12C inhibitor
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
PFS per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to Approximately 3 Years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to Approximately 5 Years
Objective Response Rate (ORR) per RECIST v1.1 | Up to Approximately 5 Years
Objective Response (OR) per RECIST v1.1 | Up to Approximately 5 Years
Duration of Response (DOR) per RECIST v1.1 | Up to Approximately 5 Years
Disease Control Rate (DCR) per RECIST v1.1 | Up to Approximately 5 Years
Time to Response (TTR) per RECIST v1.1 | Up to Approximately 5 Years
Depth of Response per RECIST v1.1 | Up to Approximately 5 Years
  Depth of response is measured as the percentage of tumor shrinkage calculated as the best percentage change from baseline in lesion sum diameters.
Time to Early Tumor Shrinkage (ETS) per RECIST v1.1 | Up to Approximately 5 Years
PFS Based on Investigator's Assessment per RECIST v1.1 | Up to Approximately 5 Years
ORR Based on Investigator's Assessment per RECIST v1.1 | Up to Approximately 5 Years
DOR Based on Investigator's Assessment per RECIST v1.1 | Up to Approximately 5 Years
DCR Based on Investigator's Assessment per RECIST v1.1 | Up to Approximately 5 Years
TTR Based on Investigator's Assessment per RECIST v1.1 | Up to Approximately 5 Years
Depth of Response Based on Investigator's Assessment per RECIST v1.1 | Up to Approximately 5 Years
Time to ETS Based on Investigator's Assessment per RECIST v1.1 | Up to Approximately 5 Years
Number of Participants Experiencing Adverse Events (AEs) | Up to Approximately 5 Years
  An AE is defined as any untoward medical occurrence in participant or clinical investigation subject administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment. A serious AE is defined as any AE that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect or important medical events that do not meet the preceding criteria but based on appropriate medical judgment may jeopardize the patient or may require medical or surgical intervention to prevent any of the outcomes listed above.
Pre-dose (Ctrough) Concentrations of Sotorasib | Day 1 (pre-dose) to week 4 (post dose) on cycle 2 (one cycle = 28 days)
Maximum Plasma Concentration (Cmax) of Sotorasib | Day 1 (pre-dose) to week 4 (post dose) on cycle 2 (one cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (282):
- United States (26):
  - Ironwood Cancer and Research Centers Scottsdale, Chandler, Arizona
  - Providence Saint Jude Medical Center, Fullerton, California
  - City of Hope National Medical Center, Long Beach, California
  - Cancer and Blood Research Center, LLC, Los Alamitos, California
  - California Research Institute, Los Angeles, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Cancer Specialists of North Florida - Southpoint, Jacksonville, Florida
  - D and H Cancer Research Center, Margate, Florida
  - Mid Florida Hematology and Oncology Centers PA, Orange City, Florida
  - Boca Raton Clinical Research Medical Center Inc, Plantation, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Insight Research Institute, Chicago, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Pikeville Medical Center, Pikeville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Saint Louis Cancer Care West County, Bridgeton, Missouri
  - Minniti Center for Medical Oncology and Hematology, Mickleton, New Jersey
  - Duke Cancer Center, Durham, North Carolina
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - Tennessee Oncology PLLC - Chattanooga, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Argentina (13):
  - Hospital Universitario Fundacion Favaloro, CABA, Buenos Aires
  - Instituto Argentino de Diagnóstico y Tratamiento, CABA, Buenos Aires
  - Investigaciones Clinicas Moleculares - Centro de Endocrinologia y Diabetes Dr Raul Gutman SRL, CABA, Buenos Aires
  - Cemic, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Sanatorio Británico de Rosario, La Plata, Buenos Aires
  - Instituto de Investigaciones clinicas de Mar del Plata, Mar del Plata, Buenos Aires
  - Hospital Italiano de Córdoba, Córdoba, Córdoba Province
  - Sanatorio Allende, Córdoba, Córdoba Province
  - Clinica Universitaria Privada Reina Fabiola, Córdoba, Córdoba Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Exelsus Oncologia Clinica, San Miguel de Tucumán, Tucumán Province
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Centro Oncologico Riojano Integral, La Rioja
- Australia (6):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Toowoomba Hospital, Toowoomba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Austin Health, Austin Hospital, Heidelberg, Victoria
- Austria (5):
  - Medizinische Universitaet Graz, Graz
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Landeskrankenhaus Feldkirch, Rankweil
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Krankenhaus Wiener Neustadt, Wiener Neustadt
- Belgium (8):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Grand Hôpital de Charleroi - Site des Viviers, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Algemeen Ziekenhuis Sint Maarten-Emmaus vzw, Mechelen
  - AZ Delta Campus Rumbeke, Roeselare
  - Vitaz campus Sint-Niklaas Moerland, Sint-Niklaas
- Brazil (16):
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Sirio Libanes Brasilia, Brasília, Federal District
  - Vencer e Oncoclinica, Teresina, Piauí
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Oncosite Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Associação Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundacao pio xII Barretos, Barretos, São Paulo
  - Oncoclinicas Belo Horizonte, Barretos, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Fundacao Antonio Prudente AC Camargo Cancer Center, São Paulo, São Paulo
  - Oncologia Rede D Or, São Paulo, São Paulo
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto Cancer Sao Paulo Icesp, São Paulo
  - Instituto Brasileiro de Controle do Cancer Ibcc, São Paulo
- Bulgaria (5):
  - Specialized Hospital for Active Treatment of Oncology - Haskovo EOOD, Haskovo
  - Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv
  - Complex Oncology Center Plovdiv EOOD, Plovdiv
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - William Osler Health System - Brampton Civic Hospital, Brampton, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Chile (8):
  - James Lind Centro de Investigacion del Cancer, Temuco, Cautín
  - Centro de investigacion y desarrollo oncolgico Spa, Temuco, Cautín
  - Enroll SpA, Providencia, Santiago Metropolitan
  - Clinica Redsalud Vitacura, Instituto del Cancer, Vitacura, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez, Santiago
  - Centro de oncologia de precision Spa, Santiago
  - Biocinetic servicios medicos limitada, Santiago
  - Clinical Research Chile SpA, Valdivia
- Colombia (6):
  - Servicios de Salud Ips Suramericana Sas - Ips Sura Industriales, Medellín, Antioquia
  - Institucion Prestadora de Servicios de Salud Sociedad Médica Rionegro SA Somer SA, Rionegro, Antioquia
  - Instituto Nacional de Cancerologia, Bogota, Cundinamarca
  - Centro de Tratamiento e Investigación sobre Cancer Luis Carlos Sarmiento Angulo Ctic, Bogotá, Cundinamarca
  - Instituto Medico de Alta Tecnologia sas - Imat sas, Montería, Departamento de Córdoba
  - Fundacion Oftalmologica de Santander - Foscal, Floridablanca, Santander Department
- Czechia (6):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
  - Fakultni nemocnice Bulovka, Prague
- Denmark (4):
  - Aalborg Sygehus, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense C
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (16):
  - Centre Hospitalier Universitaire de Clermont Ferrand - Hopital Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Dijon - Hopital du Bocage, Dijon
  - Hopital Prive Jean Mermoz, Lyon
  - Institut regional du Cancer Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint Louis, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hopital Robert Debre, Reims
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Institut de Cancerologie de l Ouest Rene Gauducheau, Saint-Herblain
  - Centre Hospitalier Universitaire Nord de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
- Germany (10):
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - UCT Universitaeres Zentrum fuer Tumorerkrankungen Frankfurt, Frankfurt am Main
  - Haematologisch Onkologische Praxis Eppendorf, Hamburg
  - Regional Kliniken Holding Klinikum Ludwigsburg, Ludwigsburg
  - Klinikum der LMU Muenchen, München
  - Universitaetsklinikum Ulm, Ulm
  - Klinikum der Stadt Wolfsburg, Wolfsburg
- Greece (10):
  - General Hospital Evangelismos, Athens
  - Agios Savvas Anticancer Hospital, Athens
  - Aretaieio Hospital, Athens
  - Hygeia Hospital, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Larissa, Larissa
  - Metaxa Anticancer Hospital, Piraeus
  - Genesis Mikti Idiotiki Gynaikas A.E. Maieutiki Gynaikologiki Cheirourgiki, Pylaia, Thessaloniki
  - Saint Lukes Hospital SA, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Princess Margaret Hospital, Kowloon
  - Tuen Mun Hospital, New Territories
- Hungary (6):
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaz, Nyíregyháza
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Italy (19):
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Ente Ospedaliero IRCCS Saverio De Bellis, Castellana Grotte
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola FC
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Specialistica dei Colli Monaldi, Napoli
  - Istituto Nazionale dei Tumori IRCCS Fondazione Giovanni Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
  - Azienda Sanitaria Territoriale Pesaro Urbino - Presidio San Salvatore Muraglia, Pesaro
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Unità Sanitaria Locale della Romagna Presidio ospedaliero di Ravenna, Ravenna
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Fondazione IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Sanitaria Universitaria Friuli Centrale Presidio Ospedaliero Santa Maria della Misericordia, Udine
  - Azienda Ospedaliera Universitaria Integrata di Verona Ospedale Civile Maggiore Borgo Trento, Verona
- Japan (19):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka
  - The University of Osaka Hospital, Suita-shi, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Tokushima University Hospital, Tokushima, Tokushima
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Mexico (4):
  - Centro Especializado en Investigacion y Tratamiento Oncologicos SC, Benito Juárez, Mexico City
  - Health Pharma Professional Research SA de CV, Mexico City, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
- Netherlands (5):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek, Amsterdam
  - Albert Schweitzer Ziekenhuis, Locatie Dordwijk, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (8):
  - Szpitale Pomorskie spolka z ograniczona odpowiedzialnoscia, Gdynia
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej w Kielcach, Kielce
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - SPZOZ Opolskie Centrum Onkologii imienia prof Tadeusza Koszarowskiego w Opolu, Opole
  - Wielkopolskie Centrum Onkologii imienia Marii Sklodowskiej-Curie, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Warsaw
- Portugal (9):
  - Unidade Local de Saude de Almada-Seixal, EPE - Hospital Garcia de Orta, Almada
  - Instituto Portugues de Oncologia de Coimbra Francisco Gentil, EPE, Coimbra
  - Unidade Local de Saude de Coimbra, EPE, Coimbra
  - Hospital Cuf Tejo, Lisbon
  - Fundacao Champalimaud, Lisbon
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Unidade Local de Saude de Entre Douro e Vouga, EPE - Hospital de Sao Sebastiao, Santa Maria da Feira
- Romania (7):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic Prof Dr Alexandru Trestioreanu Bucuresti, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - SC Oncomed SRL, Timișoara
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (20):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Institut Catala d Oncologia Badalona Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Institut Catala d Oncologia Hospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Complexo Hospitalario Universitario de Ourense, Ourense, Galicia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Elche, Elche, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Soedersjukhuset, Stockholm, Sweden
- Universitaetsspital Zuerich, Zurich, Switzerland
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Siriraj Hospital, Bangkok, Thailand
- Turkey (Türkiye) (13):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi, Edirne
  - Bezmialem Vakif Universitesi Hastanesi, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Acibadem Altunizade Hastanesi, Istanbul
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Necmettin Erbakan Universitesi Tip Fakultesi Hastanesi, Konya
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
- United Kingdom (10):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital, London
  - Guys Hospital, London
  - Royal Marsden Hospital, London
  - Sarah Cannon Research Institute UK, London
  - Maidstone Hospital, Maidstone
  - Mount Vernon Cancer Centre, Northwood
  - Weston Park Hospital, Sheffield
  - Royal Marsden Hospital - Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com